CLINICAL TRIAL: NCT03518866
Title: A Feasibility Study to Monitor Post Discharge Activity of Patient Recovery After Knee Replacement Surgery
Brief Title: Patient Recovery After Knee Replacement Surgery
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Bev Hoddell (Other Government)
Collaborators: Open University (Other)
Responsible Party: Sponsor-Investigator, Bev Hoddell, Academic Research Coordinator, Milton Keynes University Hospital NHS Foundation Trust
Organization: Milton Keynes University Hospital NHS Foundation Trust (Other Government)
Other Study IDs: 14-MK-002
Record Dates: First submitted 2017-09-11; First posted 2018-05-08 (Actual); Last update posted 2018-05-08 (Actual); Status verified 2018-04

CONDITIONS: Total Knee Replacement

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This main objective of this feasibility study is to begin to quantify the relationship between patient activity levels following knee replacement surgery and outcomes.

DETAILED DESCRIPTION:
This main objective of this feasibility study is to begin to quantify the relationship between patient activity levels following knee replacement surgery and outcomes.

Primary Aims The primary objective of this study is to compare step count and activity levels with key outcome measures - including pain scores and painkiller usage - to determine whether more active people have better recovery.

ELIGIBILITY:
Inclusion Criteria:

* Adult

* Must be able to converse and understand English
* The participants must be selected for for single full knee replacement surgery at Milton Keynes University Hospital
* The participant must have access to a computer at home or be willing to plug a synchronization box into their broadband router
* The participants must have access to a valid email address or be able to create one for the purpose of this study (this may belong to a spouse, partner, friend or relative) or have access to a mobile phone able to receive SMS (text) messages

Exclusion Criteria:

* Insufficient language skills to understand the study procedures
* Cognitive impairment
* Medical conditions (e.g., severe neurological disorder, acute cancer, psychiatric disorder, acute infections) that prevent participation in the study
* Wheelchair user
* Significant lower limb arthritic joints
* Severe mobility limitation due to central or peripheral respiratory dysfunction
* Severe mobility limitation due to central or peripheral nervous system disorders
* Severe mobility limitation due to spinal condition
* Severe mobility limitation due to musculoskeletal disabilities
* Rheumatoid arthritis due to joint pain in both upper and lower limbs
* Amputee
* Dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults undergoing elective single total knee replacement surgery at Milton Keynes University Hospital under the care of the principal investigator with no other relevant co-morbidities.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2015-07-21 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in mean weekly step count between pre surgery and 6 weeks post surgery. | 7 weeks
  Daily activity level of participant as measured by step count automatically on commercial step counter at one minute granularity from up to one week before surgery up to 6 weeks post surgery. Step count data for days which are deemed non compliant (not wearing device long enough) will be ignored. Total average daily step count (for compliant days) each week will be reported.
  The outcome measure we plan to use will be the mean daily step count from the 6th week post op. The baseline will be the mean step count from the 1 week prior to surgery.
Mean Daily Pain Score over 6 weeks following surgery | 6 weeks
  Participants will be asked to record their NRS-11 (Numeric Rating Scale) pain level in the morning, afternoon and evening daily in a paper diary for six weeks after surgery. NRS-11 is an integer scale from 0-10 with 0 representing no pain and 10 representing worst pain possible.
  The outcome measure will be the mean pain score from the 6 week post op period.
Mean weekly Oxford Knee Score for 6 weeks following surgery. | 6 weeks
  For the 6 weeks following surgery, at the end of each week patients will be asked to fill in the 12 question Oxford Knee Score (OKS) questionnaire which will result in an integer score from 0-48 for each week.
  The outcome measure will be the mean OKS over the 6 week post op period.
The OKS (Oxford Knee Score) at 6 months post surgery | 6 months
  Routine physiotherapy review appointment 6 months post surgery. OKS is collected and uploaded to standard hospital outcomes database.
The OKS (Oxford Knee Score) at 12 months post surgery | 12 months
  Routine physiotherapy review appointment 12 months post surgery. OKS is collected and uploaded to standard hospital outcomes database.
The Pain score at 6 months post surgery | 6 months
  Routine physiotherapy review appointment 6 months post surgery. Pain score is collected and uploaded to standard hospital outcomes database.
The Pain score at 12 months post surgery | 12 months
  Routine physiotherapy review appointment 12 months post surgery. Pain score is collected and uploaded to standard hospital outcomes database.

CONTACTS AND LOCATIONS:
Overall Officials: Blaine Price, Study Chair — Open University
Locations (1):
- Milton Keynes University Hospital NHS Foundation Trust, Milton Keynes, Bucks, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised raw participant data for basic demographics, surgery date, daily step count, pain scores, Oxford Knee scores will be shared on the institutional open data archive.
Supporting Information: Study Protocol
Time Frame: Raw data will be published on the institutional open data archive when the first publication is submitted for review and available for 10 years. Submission is anticipated in mid to late 2018.
Access Criteria: Open access as patient data anonymised.

REFERENCES:
- [Derived] Kelly R, Jones S, Price B, Katz D, McCormick C, Pearce O. Measuring Daily Compliance With Physical Activity Tracking in Ambulatory Surgery Patients: Comparative Analysis of Five Compliance Criteria. JMIR Mhealth Uhealth. 2021 Jan 26;9(1):e22846. doi: 10.2196/22846. PMID 33496677